CLINICAL TRIAL: NCT07378540
Title: Evaluation Of Periodontal Status In Gastritis Patients With Clinical And Microbiological Parameters
Brief Title: Evaluation of Microbial Status in Gastritis Patients in Different Periodontal Conditions
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Veli Özgen Öztürk, Principal Investigator, Aydin Adnan Menderes University
Other Study IDs: BAP-24004
Record Dates: First submitted 2026-01-16; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2024-03

CONDITIONS: Periodontal Diseases; Gastritis
Keywords: gastritis; microbiome; metagenomic analysis; dysbiosis
MeSH Terms: conditions — Periodontal Diseases; Gastritis; Dysbiosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastritis: Patients diagnosed with gastritis via endoscopic method and without other systemic diseases
  Interventions: Other: saliva collection
- Systemically healthy: Patients without any systemic disease
  Interventions: Other: saliva collection

INTERVENTIONS:
Other: saliva collection — collecting unstimulated saliva

SUMMARY:
The aim of this study to evaluate the microbial profile in gastritis and healthy patients in different periodontal conditions via next generation technologies.

DETAILED DESCRIPTION:
This study aims to determine the density of bacteria associated with periodontal disease and to evaluate oral dysbiosis in gastritis patients using metagenomic analysis.

ELIGIBILITY:
Inclusion Criteria:

* no systemic diseases other than gastritis non-smoker

Exclusion Criteria:

* Participants who took regular medications that could affect of periodontal tissue or oral microbiome pregnancy or lactation Patients who received periodontal treatment within the last 6 months

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: older than 18 years, have no systemic disease other than gastritis, non smoker participants
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Salivary microbial profile | 1 month
  To compare the oral flora profiles of the study groups, a microbiome-based next-generation sequencing approach targeting the 16S rRNA gene was employed. In this metagenomic study, following DNA extraction, phylogenetic classification was performed using the V3-V4 hypervariable regions of the 16S rRNA gene. Using the obtained data, total bacterial diversity and density were compared through alpha and beta diversity analyses. Bacterial taxa that differed between the groups were identified using LEfSe analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes University, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided